CLINICAL TRIAL: NCT03266770
Title: The RELIEF™ Ureteral Stent - Assessment of Retrograde Urinary Reflux and Distal Coil Bladder Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Kyle Scarberry, MD, Assistant Professor, Urology, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-17-30
Record Dates: First submitted 2017-08-17; First posted 2017-08-30 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Ureteral Obstruction
Keywords: ureteral stent
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- RELIEF stent placement (Other): After meeting the inclusion criteria and being consented, patients will have the RELIEF stent inserted in the ureter during cystoscopy per standard of care for ureteral stent placement.
  Interventions: Device: RELIEF Stent

INTERVENTIONS:
Device: RELIEF Stent — The RELIEF stent will be placed under cystoscopy. The stent with pusher will be placed over the guidewire and inserted. The pusher will be positioned, the guidewire will be removed, and the pusher will be retracted. The position of the stent will be confirmed by x-ray (C-arm).

SUMMARY:
Traditional ureteral stents are commonly used in renal and ureteral procedures, and their use is associated with many morbidities which can affect patients' quality of life. However, replacement of the distal portion of the stent with a thin material may reduce bladder irritative symptoms and allow the ureterovesical junction to coapt---thereby, reducing urinary reflux. The hypothesis is that the RELIEF stent will offer the same function of traditional ureteral stents with the added benefits of minimizing urinary reflux and reducing irritative bladder symptoms.

DETAILED DESCRIPTION:
Traditional ureteral stents are commonly used in practice to relieve renal obstruction or as a scaffold to promote healing after endoscopic or open/ laparoscopic surgeries involving the ureter. However, there are many morbidities associated with stent placement either due to bladder irritation or backflow of urine to the kidney. The most commonly reported symptoms include urgency, urinary frequency, dysuria, incontinence, hematuria, suprapubic discomfort, and fever due to urinary tract infections and flank pain, which can occur in up to 80% of stented patients. Sometimes, the symptoms are poorly tolerated and can negatively affect patients' quality of life. Shao et al have studied the relationship between bladder filling and the renal pelvic pressure (RPP) in stented patients, which revealed that RPP increased mildly during bladder filling and increased dramatically during voiding, indicating urinary reflux, and thus encouraging early stent removal. Another study showed that patients with stents whose distal coils cross the midline are at higher risk of post-stenting morbidities. Replacement of the distal portion of the ureteral stent with a thin material may reduce bladder irritative symptoms and allow the ureterovesical junction to coapt, thereby eliminating urinary reflux.

The Ureteral Stent Company, LLC (USC) is developing the RELIEF™ Ureteral Stent, a single use, disposable ureteral stent (US) device that will provide the traditional function of allowing the passage of urine from the kidney to the bladder with new design enhancements to improve patient care:

* A low-profile tether through the intramural ureter segment, minimizing the potential of urinary reflux
* Polymeric solid distal coil that minimizes the potential for coil positioning on the trigone, reducing the potential for associated bladder spasms and pain.

It is hypothesized that the RELIEF stent will offer the same function of traditional ureteral stents with the added benefits of minimizing the urinary reflux and reducing irritative bladder symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ureteral stone of 5-25 mm measured on plain abdomen X-ray KUB (Kidney Ureter Bladder) or CT (computed tomography).
* Upper or middle third ureteral stricture.

Exclusion Criteria:

* Patients with distal ureteral obstruction
* Patients with urinary reflux
* Patients requiring bilateral surgical stone management procedure
* Intraoperative exclusion: Based on the urologist's discretion, if trauma has been induced to the distal ureter due to ureteroscopy maneuvers, these patients will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Scarberry, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Chew BH, Knudsen BE, Denstedt JD. The use of stents in contemporary urology. Curr Opin Urol. 2004 Mar;14(2):111-5. doi: 10.1097/00042307-200403000-00011. PMID 15075840
- [Background] Joshi HB, Okeke A, Newns N, Keeley FX Jr, Timoney AG. Characterization of urinary symptoms in patients with ureteral stents. Urology. 2002 Apr;59(4):511-6. doi: 10.1016/s0090-4295(01)01644-2. PMID 11927301
- [Background] Chambade D, Thibault F, Niang L, Lakmichi MA, Gattegno B, Thibault P, Traxer O. [Study of the safety of double J ureteric stents]. Prog Urol. 2006 Sep;16(4):445-9. French. PMID 17069037
- [Background] Shao Y, Shen ZJ, Zhuo J, Liu HT, Yu SQ, Xia SJ. The influence of ureteral stent on renal pelvic pressure in vivo. Urol Res. 2009 Aug;37(4):221-5. doi: 10.1007/s00240-009-0199-z. Epub 2009 Jun 10. PMID 19513705
- [Background] Giannarini G, Keeley FX Jr, Valent F, Manassero F, Mogorovich A, Autorino R, Selli C. Predictors of morbidity in patients with indwelling ureteric stents: results of a prospective study using the validated Ureteric Stent Symptoms Questionnaire. BJU Int. 2011 Feb;107(4):648-54. doi: 10.1111/j.1464-410X.2010.09482.x. PMID 20590539
- [Background] Krebs A, Deane LA, Borin JF, Edwards RA, Sala LG, Khan F, Abdelshehid C, McDougall EM, Clayman RV. The 'buoy' stent: evaluation of a prototype indwelling ureteric stent in a porcine model. BJU Int. 2009 Jul;104(1):88-92. doi: 10.1111/j.1464-410X.2008.08338.x. Epub 2009 Jan 14. PMID 19154469

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RELIEF Stent Placement
Started | 24
Completed | 19
Not Completed | 5
Not completed — Physician Decision | 3
Not completed — Insufficient study supplies | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | RELIEF Stent Placement
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Bladder Irritation Symptoms (e.g. Frequency, Urgency, Nocturia, Urine Leakage...) Associated With the RELIEF Stent.
Description: Ureteral Stent Symptoms Questionnaire (USSQ Scale) will be used to evaluate bladder irritation symptoms at 24 hours post op. The USSQ produces a score of 19 to 220 or above where a higher score means more or worse symptoms.
Time Frame: 24 hours post op
Population: Only patients with complete responses to the USSQ at 1-day following RELIEF Stent placement were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | RELIEF Stent Placement
Number analyzed (Participants) | 16
Units on a scale | 51.95 (18.2)

2. Primary Outcome: Change in Loin Pain Scores From Baseline
Description: The 1-10 Visual Analog Scale part of the Ureteral Stent Symptoms Questionnaire (USSQ Scale) will be used to evaluate the change of loin pain from baseline. The VAS produces a score of 0 to 10 where a higher score means more or worse symptoms.
Time Frame: Baseline, Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RELIEF Stent Placement
Number analyzed (Participants) | 9
units on a scale
  Baseline | 1.33 (2.69)
  30 days | 1.22 (2.11)
Statistical Analysis 1: Comparison: RELIEF Stent Placement; Test type: Superiority; p = 0.83, t-test, 2 sided; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-1.07 to 1.29]

3. Secondary Outcome: Incidence of RELIEF Stent-Related Adverse Events
Description: Assessment of adverse events (incidence, relationship to device, severity) attributed to the RELIEF stent compared to established adverse event rates from published clinical studies and FDA reported events of conventional ureteral stents.
Time Frame: 0-30 days.
Measure: Number; unit: Adverse Events
Arm/Group | RELIEF Stent Placement
Number analyzed (Participants) | 19
Adverse Events | 3

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | RELIEF Stent Placement
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RELIEF Stent Placement (N=24)
Pain (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT03266770/Prot_001.pdf